CLINICAL TRIAL: NCT04464564
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 (Deudextromethorphan Hydrobromide [d6-DM]/Quinidine Sulfate [Q]) for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of AVP-786 for the Treatment of Agitation in Patients With Dementia of the Alzheimer's Type
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The AVP-786 program was discontinued, the recruitment was stopped and all participants are no longer being examined or receiving intervention.
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-AVP-786-307; 2020-000799-39 (EudraCT Number); 2023-504991-31-00 (EU CTIS Number)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Agitation in Patients With Dementia of the Alzheimer's Type
Keywords: Agitation; Dementia of the Alzheimer's type; Alzheimer's disease; AVP-786; Deudextromethorphan hydrobromide; Quinidine sulfate
MeSH Terms: conditions — Psychomotor Agitation; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants who were enrolled in 1-week double-blind placebo lead-in Period A, were then randomized to receive AVP-786 matching placebo capsules, twice a day, for 11 weeks in Period B.
  Interventions: Drug: Placebo
- AVP-786-18 (Experimental): Participants who were enrolled in 1-week double-blind placebo lead-in Period A, were then randomized to receive AVP-786-18 (d6-DM 18 milligrams (mg)/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
  Interventions: Drug: AVP-786
- AVP-786-42.63 (Experimental): Participants who were enrolled in 1-week double-blind placebo lead-in Period A, were then randomized to receive AVP-786-42.63 (d6-DM 42.63 mg/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
  Interventions: Drug: AVP-786

INTERVENTIONS:
Drug: AVP-786 — oral capsules
  Arms: AVP-786-18; AVP-786-42.63
Drug: Placebo — oral capsules
  Arms: Placebo

SUMMARY:
This study was conducted to evaluate the efficacy, safety, and tolerability of AVP-786 (deudextromethorphan hydrobromide [d6-DM]/quinidine sulfate [Q]) compared to placebo for the treatment of agitation in participants with dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
Eligible participants for this study had a diagnosis of probable Alzheimer's disease (AD) and had clinically significant, moderate/severe agitation secondary to AD.

This was multicenter, randomized, double-blind, placebo-controlled study, consisting of 12 weeks of treatment. Screening occurred within 4 weeks prior to randomization. Following screening procedures for assessment of inclusion and exclusion criteria, eligible participants were randomized into the study.

241 participants were enrolled into the study.

Study medication was administered orally twice daily from Day 1 through Day 85.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of probable Alzheimer's disease according to the 2011 Neuropsychiatric Inventory Agitation/Aggression (NPI-AA) working groups criteria
* Participants with clinically significant, moderate-to-severe agitation for at least 2 weeks prior to Screening that interferes with daily routine per the Investigator's judgment
* Participants who require pharmacotherapy for the treatment of agitation per the Investigator's judgment after an evaluation of reversible factors and a course of nonpharmacological interventions
* Diagnosis of agitation must meet the International Psychogeriatric Association (IPA) provisional definition of agitation.
* Participants meeting an additional predetermined blinded eligibility criterion, which will remain blinded to the clinical study site Investigators and staff
* Participants with a reliable caregiver who is able and willing to comply with all study procedures, including adherence to administering study drug and not administering any prohibited medications during the course of the study, and who spends a minimum of 2 hours per day for 4 days per week with the participant

Exclusion Criteria:

* Participants with dementia predominantly of the non-Alzheimer's type (e.g., vascular dementia, frontotemporal dementia, Parkinson's disease, substance-induced dementia)
* Participants with symptoms of agitation that are not secondary to Alzheimer's dementia (e.g., secondary to pain, other psychiatric disorder, or delirium)
* Participants with co-existent clinically significant or unstable systemic diseases that could confound the interpretation of the safety results of the study (e.g., malignancy [except skin basal-cell carcinoma], poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, or unstable valvular heart disease)
* Participants with myasthenia gravis

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (106):
- United States (46):
  - Clinical Research Site #840-020, Phoenix, Arizona
  - Clinical Research Site #840-047, Anaheim, California
  - Clinical Research Site #840-090, Costa Mesa, California
  - Clinical Research Site #840-059, Lafayette, California
  - Clinical Research Site #840-048, Lomita, California
  - Clinical Research Site #840-095, Long Beach, California
  - Clinical Research Site #840-004, Los Angeles, California
  - Clinical Research Site #840-006, Panorama City, California
  - Clinical Research Site, San Diego, California
  - Clinical Research Site #840-070, Apopka, Florida
  - Clinical Research Site #840-055, Bradenton, Florida
  - Clinical Research Site #840-096, Cape Coral, Florida
  - Clinical Research Site #840-077, Clermont, Florida
  - Clinical Research Site #840-066, Coral Springs, Florida
  - Clinical Research Site #840-039, Hallandale, Florida
  - Clinical Research Site #840-089, Kissimmee, Florida
  - Clinical Research Site #840-034, Lady Lake, Florida
  - Clinical Research Site #840-037, Miami, Florida
  - Clinical Research Site #840-092, Miami, Florida
  - Clinical Research Site #840-041, Miami, Florida
  - Clinical Research Site #840-007, Miami, Florida
  - Clinical Research Site #840-103, Miami, Florida
  - Clinical Research Site #840-042, Miami, Florida
  - Clinical Research Site #840-051, Naples, Florida
  - Clinical Research Site #840-087, Orlando, Florida
  - Clinical Research Site 840-028, Pensacola, Florida
  - Clinical Research Site # 840-105, Tampa, Florida
  - Clinical Research Site #840-104, Tampa, Florida
  - Clinical Research Site #840-049, West Palm Beach, Florida
  - Clinical Research Site #840-036, Winter Park, Florida
  - Clinical Research Site #840-065, Atlanta, Georgia
  - Clinical Research Site #840-030, Chicago, Illinois
  - Clinical Research Site #840-073, Boston, Massachusetts
  - Clinical Research Site #840-014, Bloomfield Township, Michigan
  - Clinical Research Site #840-022, Detroit, Michigan
  - Clinical Research Site #840-024, O'Fallon, Missouri
  - Clinical Research Site #840-031, Buffalo, New York
  - Clinical Research Site #840-021, Manhasset, New York
  - Clinical Research Site #840-058, New Hyde Park, New York
  - Clinical Research Site #840-035, Cypress, Texas
  - Clinical Research Site #840-053, Dallas, Texas
  - Clinical Research Site #840-093, El Paso, Texas
  - Clinical Research Site #840-072, Houston, Texas
  - Clinical Research Site #840-057, Houston, Texas
  - Clinical Research Site #840-086, Mesquite, Texas
  - Clinical Research Site #840-044, Fairfax, Virginia
- Belgium (4):
  - Clinical Research Site #056-005, Alken, Limburg
  - Clinical Research Site #056-004, Brussels
  - Clinical Research Site #056-003, Leuven
  - Clinical Research Site # 056-002, Liège
- Canada (2):
  - Clinical Research Site #124-003, Kelowna, British Columbia
  - Clinical Research Site #124-008, Québec, Quebec
- Chile (6):
  - Clinical Research Site #152-007, Viña Del Mar, Santiago Metropolitan
  - Clinical Research Site #152-002, Antofagasta
  - Clinical Research Site #152-005, Independencia
  - Clinical Research Site #152-001, Santiago
  - Clinical Research Site #152-003, Santiago
  - Clinical Research Site #152-006, Santiago
- Colombia (6):
  - Clinical Research Site #170-003, Bogotá, Columbia
  - Clinical Research Site #170-002, Pereira, Columbia
  - Clinical Research Site #170-007, Floridablanca, Santander Department
  - Clinical Research Site #170-006, Bello
  - Clinical Research Site #170-001, Bogotá
  - Clinical Research Site #170-004, Bogotá
- Croatia (6):
  - Clinical Research Site #191-008, Pula, Istria County
  - Clinical Research Site# 191-006, Rijeka
  - Clinical Research Site# 191-001, Zagreb
  - Clinical Research Site #191-003, Zagreb
  - Clinical Research Site #191-005, Zagreb
  - Clinical Research Site #191-002, Zagreb
- Hungary (4):
  - Clinical Research Site #348-002, Gyöngyös, Heves County
  - Clinical Research Site #384-001, Budapest
  - Clinical Research Site #384-003, Budapest
  - Clinical Research Site #348-004, Zalaegerszeg
- Ireland (4):
  - Clinical Research Site #372-002, Cork
  - Clinical Research Site #372-003, Cork
  - Clinical Research Site #372-004, Dublin
  - Clinical Research Site #372-001, Dublin
- Mexico (8):
  - Clinical Research Site # 484-004, Mexico City
  - Clinical Research Site #484-008, Mérida
  - Clinical Research Site #484-006, Monterrey
  - Clinical Research Site #484-005, Monterrey
  - Clinical Research Site # 484-003, Monterrey
  - Clinical Research Site #484-010, Saltillo
  - Clinical Research Site # 484-002, Sinaloa
  - Clinical Research Site #484-009, Tlalnepantla
- Clinical Trial Site #528-001, Amsterdam, Netherlands
- Slovakia (7):
  - Clinical Research Site #703-009, Dubnica Nad Váhom, Bratislava Region
  - Clinical Research Site #703-104, Rimavská Sobota, Sobota
  - Clinical Research Site #703-006, Banská Bystrica
  - Clinical Research Site #703-002, Bardejov
  - Clinical Research Site #703-005, Košice
  - Clinical Research Site #703-003, Trenčín
  - Clinical Research Site #703-001, Vranov nad Topľou
- Slovenia (6):
  - Clinical Research Site #705-006, Murska Sobota, Brezovica
  - Clinical Research Site #705-004, Begunje na Gorenjskem
  - Clinical Research Site #705-003, Ljubljana
  - Clinical Research Site #705-002, Ljubljana
  - Clinical Research Site #705-005, Maribor
  - Clinical Research Site #705-001, Nova Gorica
- Spain (6):
  - Clinical Research Site #724-013, Seville, Andalusia
  - Clinical Research Site #724-011, Palma de Mallorca, Balearic Islands
  - Clinical Research Site #724-012, Alicante, Valenciana, Comunitat
  - Clinical Research Site # 724-007, Coslada
  - Clinical Research Site #724-009, Madrid
  - Clinical Research Site #724-006, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at clinical sites in the North America, Latin America and Europe from 11 September 2020 to 28 June 2024.
Pre-assignment Details: A total of 742 participants were screened for the study, of which 241 participants were enrolled and treated with placebo in a 1-week double-blind placebo lead-in period (period A). A total of 236 participants were then randomized to receive AVP-786 (deudextromethorphan hydrobromide [d6-DM]/quinidine sulfate [Q]) or placebo in the 11-week randomization period (period B).
Groups:
- All Enrolled: Participants received AVP-786 matching placebo capsules, twice a day, for 1 week in Period A.
- AVP-786-18: Participants who were enrolled in 1-week double-blind placebo lead-in Period A, were then randomized to receive AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
Period: Period A (Placebo lead-in)
Arm/Group | All Enrolled | Placebo | AVP-786-18 | AVP-786-42.63
Started | 241 | 0 | 0 | 0
Completed | 236 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0
Not completed — Other | 5 | 0 | 0 | 0
Period: Period B (Randomization Period)
Arm/Group | All Enrolled | Placebo | AVP-786-18 | AVP-786-42.63
Started | 0 (236 participants who completed Period A, were randomized to receive Placebo, AVP-786-18, and AVP-786-42.63 in Period B.) | 76 (Out of 236 participants who completed Period A, 76 were randomized to receive Placebo in Period B.) | 83 (Out of 236 participants who completed Period A, 83 were randomized to receive AVP-786-18 in Period B.) | 77 (Out of 236 participants who completed Period A, 77 were randomized to receive AVP-786-42.63 in Period B.)
Safety Population | 0 | 76 | 83 | 77
Completed | 0 | 56 | 61 | 52
Not Completed | 0 | 20 | 22 | 25
Not completed — Adverse Event | 0 | 1 | 2 | 8
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Study Subject Withdrawal by Parent or Guardian | 0 | 3 | 3 | 5
Not completed — Study Terminated by Sponsor | 0 | 10 | 10 | 7
Not completed — Withdrawal by Subject | 0 | 2 | 4 | 1
Not completed — Reason not Specified | 0 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants who were randomized in the double-blind period B of the study.
Groups:
- Placebo: Participants were enrolled in 1-week double-blind placebo lead-in Period A, and were then randomized to receive AVP-786 matching placebo capsules, twice a day, for 11 weeks in Period B.
- AVP-786-18: Participants were enrolled in 1-week double-blind placebo lead-in Period A, and were then randomized to receive AVP-786-18 (d6-DM 18 mg/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
- AVP-786-42.63: Participants were enrolled in 1-week double-blind placebo lead-in Period A, and were then randomized to receive AVP-786-42.63 (d6-DM 42.63 mg/Q 4.9 mg) capsules, twice a day, for 11 weeks in Period B.
- Total: Total of all reporting groups
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63 | Total
Number analyzed (Participants) | 76 | 83 | 77 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (7.27) | 76.4 (7.50) | 76.5 (7.43) | 76.0 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 49 | 55 | 146
  Male | 34 | 34 | 22 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 60 | 62 | 57 | 179
  Race: Black or African American | 8 | 3 | 4 | 15
  Race: Asian | 0 | 1 | 0 | 1
  Race: American Indian or Alaska Native | 5 | 9 | 8 | 22
  Race: Other | 3 | 8 | 8 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 39 | 46 | 48 | 133
  Ethnicity: Not Hispanic or Latino | 35 | 36 | 29 | 100
  Ethnicity: Other | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From the End of Period A (Week 1) to Week 10 in the Cohen-Mansfield Agitation Inventory (CMAI) Composite Score
Description: The CMAI is used to assess the frequency of manifestations of agitated behaviors in elderly persons. It consists of 29 agitated behaviors that are further categorized into distinct agitation syndromes, also known as CMAI factors of agitation. These distinct agitation syndromes include aggressive behavior, physically nonaggressive behavior, and verbally agitated behavior. Each of the 29 items is rated on a 7-point scale of frequency (1 = never, 2 = less than once a week but still occurring, 3 = once or twice a week, 4 = several times a week, 5 = once or twice a day, 6 = several times a day, 7 = several times an hour). The ratings are based on the 2 weeks preceding assessment of the CMAI. Higher scores indicate higher frequency of agitated behaviours while lower scores indicate lower frequency of agitated behaviours.
Time Frame: Week 1 to Week 10
Population: Due to discontinuation of development of the AVP-786 compound, no data was collected and analyzed as planned for this pre-specified primary efficacy outcome measure as noted in the SAP. Only safety data was collected and analyzed
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) and Serious TEAE
Description: An adverse event (AE) is any untoward medical occurrence or unintended change (eg, physical, psychological, or behavioral), including inter-current illness, that does not necessarily have a causal relationship with the study treatment. A serious adverse event (SAE) is any AE occurring at any dose that results in death, life-threatening experience, persistent or significant disability/incapacity, in-patient hospitalization or prolongation of hospitalization or congenital anomaly/birth defect. TEAEs are all AEs (including serious and non-serious) which started after start of double-blind study drug treatment; or if the event was continuous from baseline and was worsening, serious, study drug related, or resulted in death, discontinuation, interruption or reduction of study therapy.
Time Frame: From randomization (Week 2) up to 30 days after last dose of study drug (Up to Week 16)
Population: Safety population included of all participants who were randomized in the double-blind period B of this study, and took at least one dose of double-blind, randomized study medication. As pre-specified in the Statistical Analysis Plan (SAP), safety data was planned to be collected only for the participants who were randomized in the double-blind period B of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63
Number analyzed (Participants) | 76 | 83 | 77
Participants
  TEAEs | 25 | 38 | 34
  Serious TEAEs | 4 | 5 | 5

3. Secondary Outcome: Change From the End of Period A (Week 1) to Week 10 in the Clinical Global Impression of Severity of Illness (CGIS) Score, as Related to Agitation
Description: The CGIS is an observer-rated scale that measures illness severity. The CGIS-Agitation is a 7-point (1-7) scale (1 = normal, not at all ill; 7 = among the most extremely ill patients) and assesses severity of agitation in this study. Higher scores indicate severe agitation while the lower scores indicate little or no agitation.
Time Frame: Week 1 to Week 10
Population: Due to discontinuation of development of the AVP-786 compound, no data was collected and analyzed as planned for this pre-specified secondary efficacy outcome measure as noted in the SAP. Only safety data was collected and analyzed.
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization (Week 2) up to 30 days after last dose of study drug (Up to Week 16)
Description: Safety population included of all participants who were randomized in the double-blind period B of this study, and took at least one dose of double-blind, randomized study medication. As pre-specified in the SAP, safety data was planned to be collected only for the participants who were randomized in the double-blind period B of this study.
Arm/Group | Placebo | AVP-786-18 | AVP-786-42.63
All-Cause Mortality (participants affected / at risk) | 1/76 | 0/83 | 1/77
Serious Adverse Events (participants affected / at risk) | 4/76 | 5/83 | 5/77
Other Adverse Events (participants affected / at risk) | 25/76 | 38/83 | 32/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | AVP-786-18 (N=83) | AVP-786-42.63 (N=77)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | AVP-786-18 (N=83) | AVP-786-42.63 (N=77)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 4 | 1
Gait disturbance (General disorders) | 0 | 1 | 3
Oedema (General disorders) | 1 | 0 | 0
Unevaluable event (General disorders) | 0 | 1 | 1
Biliary cyst (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 1 | 2
Bacteriuria (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 5 | 4
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral rhinitis (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 7 | 9
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase abnormal (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase abnormal (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Heart rate decreased (Investigations) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 0
Oesophagogastroduodenoscopy (Investigations) | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1
Akinesia (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 4 | 3 | 5
Dyslalia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 2
Hypersomnia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 4
Tremor (Nervous system disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Behaviour disorder (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Enuresis (Psychiatric disorders) | 1 | 0 | 0
Hypnopompic hallucination (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Sleep talking (Psychiatric disorders) | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0
Hypercalciuria (Renal and urinary disorders) | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Edentulous (Social circumstances) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 3 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to discontinuation of development of the AVP-786 compound.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT04464564/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT04464564/SAP_001.pdf